CLINICAL TRIAL: NCT03245593
Title: Shared Medical Decision Making in the Prophylactic Treatment of Bipolar Disorder
Acronym: ShareD-BD
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PREPS/2016/LS-01
Record Dates: First submitted 2017-08-07; First posted 2017-08-10 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-02

CONDITIONS: Bipolar Disorder
MeSH Terms: conditions — Bipolar Disorder | interventions — Standard of Care

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Shared Decision making for care (Experimental)
  Interventions: Other: Shared-decision making process
- Standard decision making for care (Other)
  Interventions: Other: standard care

INTERVENTIONS:
Other: Shared-decision making process — Completion of the Ottawa Personal Decision Guide to help guide care with the support of online and printed material describing the therapeutic options available
  Arms: Shared Decision making for care
Other: standard care — Care of patients according to standard practice of managing patients with bipolar disorder
  Arms: Standard decision making for care

SUMMARY:
The investigators hypothesize that implementation of a shared decision making care plan for prophylactic treatment will help therapeutic adherence of bipolar patients. They also anticipate that patients treated according to a shared decision making plan will have an elevated satisfaction of their care, quality of life and functionment, as well as a lower number of relapses

ELIGIBILITY:
Inclusion Criteria:

* The patient must have given their free and informed consent and signed the consent form
* The patient must be a member or beneficiary of a health insurance plan
* The patient must be available for the 12 months of follow-up
* The patient is at least 18 years old
* Patients is suffering from bipolar disorder (I or II) according to DSM-5 criteria
* Following resolution of a mood episode (manic or depressive according to DSM-5 criteria) according to the criteria of l'International Society for Bipolar Disorder (Recovery, clinical remission of at least 4 weeks)
* Followed by at least one of the practitioner belonging to one of the participating centers
* Without comprehension problems of fluent French

Exclusion Criteria:

* The subject is participating in an interventional study, or has participated in another interventional study within the previous 3 months
* The subject is in a period of exclusion determined by a previous study
* The patient is under safeguard of justice or state guardianship
* It is impossible to give the subject informed information, or the subject refuses to sign the consent
* The subject has already participated in this study
* The patient has troubles linked to the usage of severe intensive substances (such as those defined by the DMS-5)
* The patient has a revision of the initial diagnosis of bipolar disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2018-04-24 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Measure the difference of prophylactic treatment compliance between bipolar patients receiving treatment according to standard care versus a shared decision making care plan following a mood episode. | 12 months
  Clinician Rating Scale (1-7)

SECONDARY OUTCOMES:
Study the clinician-reported difference between the 2 groups in medication adherence | 3 months
  Clinician Rating Scale (1-7)
Study the clinician-reported difference between the 2 groups in medication adherence | 6 months
  Clinician Rating Scale (1-7)
Study the clinician-reported difference between the 2 groups in medication adherence | 9 months
  Clinician Rating Scale (1-7)
Study the self-reported difference between the 2 groups in medication adherence | 3 months
  Medication Adherence Rating Scale( 0-10),
Study the self-reported difference between the 2 groups in medication adherence | 6 months
  Medication Adherence Rating Scale( 0-10),
Study the self-reported difference between the 2 groups in medication adherence | 9 months
  Medication Adherence Rating Scale( 0-10),
Study the self-reported difference between the 2 groups in medication adherence | 12 months
  Medication Adherence Rating Scale( 0-10),
Clinical evaluation of the difference between the 2 groups in medication adherence | 3 months
  Plasma levels of medication for treatment of bipolar disorder, Lithium, anticonvulsants, second generation antipsychotics and antidepressants
Clinical evaluation of the difference between the 2 groups in medication adherence | 6 months
  Plasma levels of medication for treatment of bipolar disorder, Lithium, anticonvulsants, second generation antipsychotics and antidepressants
Clinical evaluation of the difference between the 2 groups in medication adherence | 9 months
  Plasma levels of medication for treatment of bipolar disorder, Lithium, anticonvulsants, second generation antipsychotics and antidepressants
Clinical evaluation of the difference between the 2 groups in medication adherence | 12 months
  Plasma levels of medication for treatment of bipolar disorder, Lithium, anticonvulsants, second generation antipsychotics and antidepressants
Compare difference in the adherence to personalized follow-up between groups | 3 months
  percentage of consultations missed
Compare difference in the adherence to personalized follow-up between groups | 6 months
  percentage of consultations missed
Compare difference in the adherence to personalized follow-up between groups | 9 months
  percentage of consultations missed
Compare difference in the adherence to personalized follow-up between groups | 12 months
  percentage of consultations missed
Compare difference in patient perceptions related to the uncertainty of the medical decisions taken between groups | 3 months
  decisional conflict scale (0-100)
Compare difference in patient perceptions related to the uncertainty of the medical decisions taken between groups | 6 months
  decisional conflict scale (0-100)
Compare difference in patient perceptions related to the uncertainty of the medical decisions taken between groups | 9 months
  decisional conflict scale (0-100)
Compare difference in patient perceptions related to the uncertainty of the medical decisions taken between groups | 12 months
  decisional conflict scale (0-100)
Compare difference in patient satisfaction concerning the therapeutic decisions taken between groups | 3 months
  adapted QSH-45: 3 questions scored 1-5
Compare difference in patient satisfaction concerning the therapeutic decisions taken between groups | 6 months
  adapted QSH-45: 3 questions scored 1-5
Compare difference in patient satisfaction concerning the therapeutic decisions taken between groups | 9 months
  adapted QSH-45: 3 questions scored 1-5
Compare difference in patient satisfaction concerning the therapeutic decisions taken between groups | 12 months
  adapted QSH-45: 3 questions scored 1-5
Compare difference in patient satisfaction concerning the decision-making process between groups | 3 months
  Adapted clinical decision making involvement and satisfaction score 3 questions scored 1-5
Compare difference in patient satisfaction concerning the decision-making process between groups | 6 months
  Adapted clinical decision making involvement and satisfaction score 3 questions scored 1-5
Compare difference in patient satisfaction concerning the decision-making process between groups | 9 months
  Adapted clinical decision making involvement and satisfaction score 3 questions scored 1-5
Compare difference in patient satisfaction concerning the decision-making process between groups | 12 months
  Adapted clinical decision making involvement and satisfaction score 3 questions scored 1-5
Compare difference in therapeutic alliance between groups | 3 months
  4-Point ordinal Alliance Scale
Compare difference in therapeutic alliance between groups | 6 months
  4-Point ordinal Alliance Scale
Compare difference in therapeutic alliance between groups | 9 months
  4-Point ordinal Alliance Scale
Compare difference in therapeutic alliance between groups | 12 months
  4-Point ordinal Alliance Scale
Compare difference in knowledge of disease and treatment necessary to making decisions between groups | 3 months
  Knowledge questionnaire: % correct answers
Compare difference in knowledge of disease and treatment necessary to making decisions between groups | 6 months
  Knowledge questionnaire: % correct answers
Compare difference in knowledge of disease and treatment necessary to making decisions between groups | 9 months
  Knowledge questionnaire: % correct answers
Compare difference in knowledge of disease and treatment necessary to making decisions between groups | 12 months
  Knowledge questionnaire: % correct answers
Compare difference in patient attitude towards the treatment between groups | 3 months
  Beliefs about Medicines Questionnaire: 18 questions 1-5
Compare difference in patient attitude towards the treatment between groups | 6 months
  Beliefs about Medicines Questionnaire: 18 questions 1-5
Compare difference in patient attitude towards the treatment between groups | 9 months
  Beliefs about Medicines Questionnaire: 18 questions 1-5
Compare difference in patient attitude towards the treatment between groups | 12 months
  Beliefs about Medicines Questionnaire: 18 questions 1-5
Compare number and duration of mood episodes between groups months | 3 months
  number of events; number of days
Compare number and duration of mood episodes between groups months | 6 months
  number of events; number of days
Compare number and duration of mood episodes between groups months | 9 months
  number of events; number of days
Compare number and duration of mood episodes between groups months | 12 months
  number of events; number of days
Compare number and duration of hospitalizations in psychiatric service between groups | 3 months
  number of events; number of days
Compare number and duration of hospitalizations in psychiatric service between groups | 6 months
  number of events; number of days
Compare number and duration of hospitalizations in psychiatric service between groups | 9 months
  number of events; number of days
Compare number and duration of hospitalizations in psychiatric service between groups | 12 months
  number of events; number of days
Compare manic symptomatology during evaluations between groups | 3 months
  Young Mania Rating Scale
Compare manic symptomatology during evaluations between groups | 6 months
  Young Mania Rating Scale
Compare manic symptomatology during evaluations between groups | 9 months
  Young Mania Rating Scale
Compare manic symptomatology during evaluations between groups | 12 months
  Young Mania Rating Scale
Compare the depressive symptomatology during evaluations between groups | 3 months
  Montgomery-Asberg Depression Rating Scale
Compare the depressive symptomatology during evaluations between groups | 6 months
  Montgomery-Asberg Depression Rating Scale
Compare the depressive symptomatology during evaluations between groups | 9 months
  Montgomery-Asberg Depression Rating Scale
Compare the depressive symptomatology during evaluations between groups | 12 months
  Montgomery-Asberg Depression Rating Scale
Compare severity and intensity of suicidal ideas between groups | 3 months
  Columbia-Suicide Severity Rating Scale
Compare severity and intensity of suicidal ideas between groups | 6 months
  Columbia-Suicide Severity Rating Scale
Compare severity and intensity of suicidal ideas between groups | 9 months
  Columbia-Suicide Severity Rating Scale
Compare severity and intensity of suicidal ideas between groups | 12 months
  Columbia-Suicide Severity Rating Scale
Compare the psychosocial functioning between groups | 3 months
  Functioning Assessment Short Test (0-72)
Compare the psychosocial functioning between groups | 6 months
  Functioning Assessment Short Test (0-72)
Compare the psychosocial functioning between groups | 9 months
  Functioning Assessment Short Test (0-72)
Compare the psychosocial functioning between groups | 12 months
  Functioning Assessment Short Test (0-72)
Compare quality of life between groups | 3 months
  WHOQOL-BREF (0-100)
Compare quality of life between groups | 6 months
  WHOQOL-BREF (0-100)
Compare quality of life between groups | 9 months
  WHOQOL-BREF (0-100)
Compare quality of life between groups | 12 months
  WHOQOL-BREF (0-100)
Compare length of consultations between groups | every consultation for 12 months
  minutes
Clinician satisfaction concerning the therapeutic decisions taken between groups | 3 months
  adapted QSH-45 doctor version 3 questions scored 1-5
Clinician satisfaction concerning the therapeutic decisions taken between groups | 6 months
  adapted QSH-45 doctor version 3 questions scored 1-5
Clinician satisfaction concerning the therapeutic decisions taken between groups | 9 months
  adapted QSH-45 doctor version 3 questions scored 1-5
Clinician satisfaction concerning the therapeutic decisions taken between groups | 12 months
  adapted QSH-45 doctor version 3 questions scored 1-5
Clinician satisfaction concerning the decision-making process between groups | 3 months
  Adapted clinical decision making involvement and satisfaction score doctor version 3: questions scored 1-5
Clinician satisfaction concerning the decision-making process between groups | 6 months
  Adapted clinical decision making involvement and satisfaction score doctor version 3: questions scored 1-5
Clinician satisfaction concerning the decision-making process between groups | 9 months
  Adapted clinical decision making involvement and satisfaction score doctor version 3: questions scored 1-5
Clinician satisfaction concerning the decision-making process between groups | 12 months
  Adapted clinical decision making involvement and satisfaction score doctor version 3: questions scored 1-5
Clinician perceptions related to the uncertainty of the medical decisions taken between groups | 3 months
  decisional conflict scale doctor version (0-100)
Clinician perceptions related to the uncertainty of the medical decisions taken between groups | 6 months
  decisional conflict scale doctor version (0-100)
Clinician perceptions related to the uncertainty of the medical decisions taken between groups | 9 months
  decisional conflict scale doctor version (0-100)
Clinician perceptions related to the uncertainty of the medical decisions taken between groups | 12 months
  decisional conflict scale doctor version (0-100)

CONTACTS AND LOCATIONS:
Overall Officials: Ludovic Samalin, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (16):
- France (16):
  - Ch Beziers, Béziers
  - CH Charles Perrens, Bordeaux
  - CH le Vinatier, Bron
  - CHU de Clermont Ferrand - Hôpital Gabriel-Montpied, Clermont-Ferrand
  - Chu Gabriel Montpied Clermont Ferrand, Clermont-Ferrand
  - CH Sainte-Marie de Clermont-Ferrand, Clermont-Ferrand
  - APHP - Centre Hospitalier Henri Mondor, Créteil
  - CHU de Grenoble - Hôpital Albert Michallon, Grenoble
  - CH Limoges, Limoges
  - APHM - Hôpital Sainte-Marguerite, Marseille
  - CHU de Montpellier - Hôpital Lapeyronie, Montpellier
  - CHU Nancy, Nancy
  - CHU Nantes, Nantes
  - Clinique des troubles thymiques, Nîmes
  - CHU Nimes, Nîmes
  - APHP - Hôpital Saint Louis-Lariboisière-Fernand-Widal, Paris

REFERENCES:
- [Derived] Samalin L, Honciuc M, Boyer L, de Chazeron I, Blanc O, Abbar M, Llorca PM. Efficacy of shared decision-making on treatment adherence of patients with bipolar disorder: a cluster randomized trial (ShareD-BD). BMC Psychiatry. 2018 Apr 13;18(1):103. doi: 10.1186/s12888-018-1686-y. PMID 29653535